CLINICAL TRIAL: NCT03245866
Title: Swiss Study on Subarachnoid Hemorrhage (Swiss-SOS)
Brief Title: Swiss Study on Subarachnoid Hemorrhage
Acronym: Swiss-SOS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: University of Bern (Other); University Hospital, Basel, Switzerland (Other); Kantonsspital Aarau (Other); Ospedale Regionale di Lugano (Other); University Hospital, Zürich (Other); Cantonal Hospital of St. Gallen (Other); University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Philippe Bijlenga, MD PhD, University Hospital, Geneva
Other Study IDs: SwissSOS_0001
Record Dates: First submitted 2015-08-23; First posted 2017-08-10 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Subarachnoid Hemorrhage; Intracranial Aneurysm
Keywords: Subarachnoid Hemorrhage; Intracranial Aneurysm; Ruptured Intracranial Aneurysm; Neurosurgery; Interventional Neuroradiology; Neurointensive Care Medicine; Switzerland
MeSH Terms: conditions — Subarachnoid Hemorrhage; Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aneurysmal Subarachnoid hemorrhage: Patients suffering from a ruptured cerebral aneurysm are included in the study.
  Interventions: Other: Observational/ no intervention

INTERVENTIONS:
Other: Observational/ no intervention

SUMMARY:
This registry was created to assess management parameters of patients treated for aneurysmal subarachnoid hemorrhage in Switzerland. All Swiss hospitals with a neurosurgery department, an intensive care unit and an interventional neuroradiology team that treat neurovascular emergencies participate in the registry. Clinical parameters are entered into a common database. This database will provide (1) a nationwide assessment of the current standard of care and (2) the outcomes for patients in Switzerland including neuropsychological assessments.

DETAILED DESCRIPTION:
Overview:

The management of aneurysmal subarachnoid hemorrhage (aSAH) in Switzerland has not been assessed on a national level to date. The investigators united all comprehensive neurovascular care centres in Switzerland to create a registry for aSAH. This registry helps collect clinical and management data from different centres and pools it in one common database. It may provide referring caregivers and healthcare providers with a critical tool to assess the quality of care in a disease which has a high socio-economic burden. Moreover, it may serve as a tool to foster scientific collaboration and address a number of remaining questions about the management of aSAH in the future. Regarding SAH, data from the federal statistics bureau of Switzerland are based strictly on ICD-10 codes provided by hospitals and show an estimate of 13 per 100,000 in a population of roughly 8 million (http://bfs.admin.ch). These numbers, however, are not referring to aneurismal SAH exclusively and thus exceed the numbers which the investigators expect to obtain. The goal is to obtain complete recruitment of SAH patients throughout Switzerland, and the goal is therefore that assessment of incidence will be performed later on.

Data management:

Data is entered into a central online database created by the Secutrial platform. This platform is provided by the University Hospital of Geneva's Clinical Research Unit. The database disposes of an audit-trail capacity. Local principal investigators are responsible for data-cross check and quality management. Source data verification is performed by investigators on site who address missing data. Regular meetings are held to discuss data patency.

The platform automatically provides a report on recruitment progress.

ELIGIBILITY:
Inclusion criteria:

- Patients admitted with a proven diagnosis of aneurysmal subarachnoid hemorrhage.

Exclusion criteria:

- Patients in whom the source of haemorrhage could not be identified (angiogram-negative SAH) or SAH with other causes than cerebral aneurysms.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted in Switzerland with a diagnosis of aneurysmal subarachnoid hemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2009-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional outcome as assessed by the modified Rankin scale | 5 years after hemorrhage
  The modified Rankin scale is used to represent the level of disability and is divided into 7 categories (0-6). The scale runs from 0-6, running from perfect health without symptoms to death.
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.

CONTACTS AND LOCATIONS:
Overall Officials: Karl Schaller, MD, Study Director — University Hospital, Geneva; Bawarjan Schatlo, MD, Principal Investigator — University Hospital, Geneva; Martin N Stienen, MD, Principal Investigator — University Hospital, Geneva; Philippe Bijlenga, MD PhD, Principal Investigator — University Hospital, Geneva
Locations (9):
- Switzerland (9):
  - Kantonsspital Aarau, Aarau, Canton of Aargau
  - Geneva University Hospital, Geneva, Canton of Geneva
  - Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - University Hospital Basel, Basel
  - University Hospital Bern, Bern
  - University Hospital Lausanne, Lausanne
  - Luzerner Kanton Spital, Lucerne
  - Ospedale Civico, Lugano
  - University Hospital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No
N/A, observational study

REFERENCES:
- [Background] Zweifel-Zehnder AE, Stienen MN, Chicherio C, Studerus-Germann A, Blasi S, Rossi S, Gutbrod K, Schmid N, Beaud V, Mondadori C, Brugger P, Sacco L, Muri R, Hildebrandt G, Fournier JY, Keller E, Regli L, Fandino J, Mariani L, Raabe A, Daniel RT, Reinert M, Robert T, Schatlo B, Bijlenga P, Schaller K, Monsch AU; Swiss SOS study group. Call for uniform neuropsychological assessment after aneurysmal subarachnoid hemorrhage: Swiss recommendations. Acta Neurochir (Wien). 2015 Sep;157(9):1449-58. doi: 10.1007/s00701-015-2480-y. Epub 2015 Jul 16. PMID 26179382
- [Result] Schatlo B, Fung C, Fathi AR, Sailer M, Winkler K, Daniel RT, Bijlenga P, Ahlborn P, Seule M, Zumofen D, Reinert M, Woernle C, Stienen M, Levivier M, Hildebrandt G, Mariani L, Bernays R, Fandino J, Raabe A, Keller E, Schaller K. Introducing a nationwide registry: the Swiss study on aneurysmal subarachnoid haemorrhage (Swiss SOS). Acta Neurochir (Wien). 2012 Dec;154(12):2173-8; discussion 2178. doi: 10.1007/s00701-012-1500-4. Epub 2012 Oct 6. PMID 23053275
- [Derived] Schatlo B, Fung C, Stienen MN, Fathi AR, Fandino J, Smoll NR, Zumofen D, Daniel RT, Burkhardt JK, Bervini D, Marbacher S, Reinert M, D Alonzo D, Ahlborn P, Mendes Pereira V, Roethlisberger M, Seule M, Kerkeni H, Remonda L, Weyerbrock A, Woernle K, Venier A, Perren F, Sailer M, Robert T, Rohde V, Schoni D, Goldberg J, Nevzati E, Diepers M, Gralla J, Z'Graggen W, Starnoni D, Woernle C, Maldaner N, Kulcsar Z, Mostaguir K, Maduri R, Eisenring C, Bernays R, Ferrari A, Dan-Ura H, Finkenstadt S, Gasche Y, Sarrafzadeh A, Jakob SM, Corniola M, Baumann F, Regli L, Levivier M, Hildebrandt G, Landolt H, Mariani L, Guzman R, Beck J, Raabe A, Keller E, Bijlenga P, Schaller K. Incidence and Outcome of Aneurysmal Subarachnoid Hemorrhage: The Swiss Study on Subarachnoid Hemorrhage (Swiss SOS). Stroke. 2021 Jan;52(1):344-347. doi: 10.1161/STROKEAHA.120.029538. Epub 2020 Dec 4. PMID 33272133
- [Derived] Stienen MN, Smoll NR, Fung C, Goldberg J, Bervini D, Maduri R, Chiappini A, Robert T, May A, Bijlenga P, Zumofen D, Roethlisberger M, Seule MA, Marbacher S, Fandino J, Schatlo B, Schaller K, Keller E, Bozinov O, Regli L; Swiss SOS Study Group. Home-Time as a Surrogate Marker for Functional Outcome After Aneurysmal Subarachnoid Hemorrhage. Stroke. 2018 Dec;49(12):3081-3084. doi: 10.1161/STROKEAHA.118.022808. PMID 30735342
- [Derived] Stienen MN, Germans M, Burkhardt JK, Neidert MC, Fung C, Bervini D, Zumofen D, Rothlisberger M, Marbacher S, Maduri R, Robert T, Seule MA, Bijlenga P, Schaller K, Fandino J, Smoll NR, Maldaner N, Finkenstadt S, Esposito G, Schatlo B, Keller E, Bozinov O, Regli L; Swiss SOS Study Group. Predictors of In-Hospital Death After Aneurysmal Subarachnoid Hemorrhage: Analysis of a Nationwide Database (Swiss SOS [Swiss Study on Aneurysmal Subarachnoid Hemorrhage]). Stroke. 2018 Feb;49(2):333-340. doi: 10.1161/STROKEAHA.117.019328. Epub 2018 Jan 15. PMID 29335333